CLINICAL TRIAL: NCT05328167
Title: Contrast-Enhanced Ultrasound for Diagnosis and Therapy of Cholangiocarcinoma
Brief Title: Contrast-Enhanced Ultrasound for the Prediction of Bile Duct Cancer Response to Radioembolization Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21F.1081; JT 19280 (Other: JeffTrial Number); R21CA259750 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (perflutren protein-type A microspheres, CEUS) (Experimental): Patients receive perflutren protein-type A microspheres IV over 10 minutes and undergo ultrasound at 1 month before TARE, 1-4 hours, 1 week, and 2 weeks post-TARE.
  Interventions: Drug: Perflutren Protein-Type A Microspheres; Procedure: Contrast-Enhanced Ultrasound

INTERVENTIONS:
Drug: Perflutren Protein-Type A Microspheres — Given IV
  Other Names: Optison
Procedure: Contrast-Enhanced Ultrasound — Undergo CEUS
  Other Names: CEUS

SUMMARY:
This phase II trial tests whether contrast-enhanced ultrasound can predict the response of bile duct cancer to targeted radiotherapy (radioembolization treatment). Contrast-enhanced ultrasound uses gas microbubbles that may provide enhancement on ultrasound. It is also possible to pop these microbubbles using ultrasound imaging. Tumors that experience popping of these microbubbles may be easier to kill with radiotherapies. Therefore, this trial may also help doctors see if ultrasound-triggered microbubble popping can improve bile duct cancer response to radiotherapy. Another purpose of this trial is to test if the pressure inside the tumor estimated through ultrasound can be used to predict the tumor response to radiotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the ability of quantitative volumetric contrast-enhanced ultrasound (CEUS) to predict non-hepatocellular carcinoma (HCC) tumor response to transarterial radioembolization (TARE) prior to therapy.

SECONDARY OBJECTIVES:

I. To characterize the safety and preliminary efficacy of using localized ultrasound contrast agent (UCA) inertial cavitation to improve ICC response to radioembolization.

II. To determine if CEUS estimated tumor perfusion and residual vascularity 7-14 days post treatment can predict ICC response to radioembolization.

III. To evaluate tumoral response using the patient's 1 month magnetic resonance imaging (MRI) (obtained clinically) and determine the accuracy of MR or computed tomography (CT) tumor evaluation at this earlier time point.

EXPLORATORY OBJECTIVE:

I. To examine the utility of subharmonic aided pressure estimation (SHAPE) to noninvasively monitor tumoral interstitial fluid pressure (IFP) and provide an early biomarker of radiotherapy response.

OUTLINE:

Patients receive perflutren protein-type A microspheres intravenously (IV) over 10 minutes and undergo ultrasound at 1 month before TARE, 1-4 hours, 1 week, and 2 weeks post-TARE.

After completion of study, patients are followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled for sub-lobar radioembolization therapy of a previously untreated intrahepatic cholangiocarcinoma greater than 1 cm but small enough to be fully visualized in the ultrasound three-dimensional (3D) volume (approximately 6 cm maximum diameter, but depth dependent)
* Be at least 18 years of age
* Be medically stable
* If a female of child-bearing age, have a negative pregnancy test prior to each ultrasound exam
* Have signed Informed Consent to participate in the study

Exclusion Criteria:

* Females who are pregnant or nursing
* Patients with recent cerebral hemorrhage
* Patients with known sensitivities to albumin, blood, or blood products
* Patients with known hypersensitivity to perflutren
* Patients with known congenital heart defects
* Patients with severe emphysema, pulmonary vasculitis, or a history of pulmonary emboli
* Patients with bilirubin levels > 2 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diagnostic (perflutren protein-type A microspheres, CEUS)
Started | 16
Completed | 14
Not Completed | 2
Not completed — Treatment cancelled prior to radioembolization | 1
Not completed — imaging not obtained for primary outcome assessment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Diagnostic (perflutren protein-type A microspheres, CEUS)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tumor Complete Response (CR)
Description: Assessed by modified RECIST (mRECIST) criteria using contrast-enhanced CT or MRI reviewed by two independent readers. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), indicated by a significant increase (at least 20%) in target lesions or the appearance of new target lesions; Stable Disease (SD) means neither the criteria for PR nor for Progressive Disease (PD) have been met.
Time Frame: assessed at 3 to 6 months post-TARE
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (perflutren protein-type A microspheres, CEUS)
Number analyzed (Participants) | 14
Participants | 7

2. Primary Outcome: Number of Participants With Tumor Partial Response (PR)
Description: as for outcome 1
Time Frame: assessed at 3 to 6 months post-TARE
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (perflutren protein-type A microspheres, CEUS)
Number analyzed (Participants) | 14
Participants | 3

3. Primary Outcome: Number of Participants With Stable Disease
Description: as for outcome 1
Time Frame: assessed at 3 to 6 months post-TARE
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (perflutren protein-type A microspheres, CEUS)
Number analyzed (Participants) | 14
Participants | 4

4. Primary Outcome: Number of Participants With Progressive Disease
Description: as for outcome 1
Time Frame: assessed at 3 to 6 months post-TARE
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic (perflutren protein-type A microspheres, CEUS)
Number analyzed (Participants) | 14
Participants | 0

ADVERSE EVENTS:
Time Frame: The PI will follow adverse events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation, up to 6 months post-baseline. At each study visit, the investigator (or designee) will inquire about the occurrence of AE/SAEs since the last visit. Events will be followed for outcome information until resolution or stabilization.
Description: Adverse events were monitored through systematic assessments including clinical observation, patient self-report, and medical record review at study visits from informed consent through 30 days after last study visit.
Arm/Group | Diagnostic (perflutren protein-type A microspheres, CEUS)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT05328167/Prot_SAP_000.pdf